CLINICAL TRIAL: NCT02294487
Title: The Immune Response Following Vaccination in Multiple Myeloma Patients: A Prospective Pilot Study
Brief Title: Study of the Immune Response After Vaccination in Multiple Myeloma Patients
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Vince Lombardi Cancer Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MMvax-pilot
Record Dates: First submitted 2014-10-21; First posted 2014-11-19 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma; Myeloma, Multiple; Myeloma-Multiple
Keywords: influenza; pneumococcal; pneumonia; vaccine; immunization; #CAImmun; Immuno-oncology; supportive care; vaccination; meningococcal; HIB
MeSH Terms: conditions — Multiple Myeloma; Influenza, Human; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects: Individuals over 50 who are going to get the seasonal flu vaccine, pneumococcal, HIB, and/or meningococcal vaccination and either have multiple myeloma or do not have multiple myeloma.

SUMMARY:
This study will collect blood samples from healthy volunteers and volunteers with multiple myeloma who are going to get the seasonal flu, pneumonia, haemophilus influenzae B (HIB), and/or meningococcus vaccines.

The main goal of the study is to start to identify differences in the immune response between multiple myeloma patients and people who don't have multiple myeloma. We hope this will provide important information about the best way and time to vaccinate multiple myeloma patients to flu, pneumonia, haemophilus influenzae B (HIB), and/or meningococcus .

DETAILED DESCRIPTION:
This study will consist of a prospective blood sample collection to gather baseline data to confirm antibody protection from vaccines in the Aurora Health Care multiple myeloma (MM) patients.

The overall goal of this study is to obtain a normative dataset for MM patients and non-MM control populations as well as determining baseline IgG levels to seasonal influenza A, influenza B, pneumococcal polysaccharide, and tetanus toxoid and confirmation of antibody protection from vaccines with assays based upon WHO standards of detection.

This is part of a series of studies designed to provide important information about the best way and time to vaccinate MM patients to flu, pneumonia, haemophilus influenzae B (HIB), and/or meningococcus and to gather additional information about MM and immune function.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or over
* planning on getting the seasonal flu and/or pneumonia vaccine as part of normal care
* have multiple myeloma, or don't have multiple myeloma and want to serve as a health control

Exclusion Criteria:

- do not meet inclusion criteria

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients and age and sex matched control subjects over 50 who are already planning to have the flu and/or pneumonia vaccine as part of normal care. The control group is important for comparison of age-adjusted changes in immune responses to vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluate composition of T cells, B cells, NK cell and monocyte populations from pre-vaccination though 24 weeks post-vaccination | 24 weeks
  Evaluate composition of T cells, B cells, NK cell and monocyte populations to identify immune suppression. Multiparameter flow cytometer will be used to evaluate T cells, B cells, and NK cell and monocyte populations using differentiation markers for the cell populations in subjects at five time points, baseline to 24 weeks.
Measure of interferon -gamma in activated T cells from pre-vaccination though 24 weeks post-vaccination | 24 weeks
  Measure of interferon -gamma in activated T cells to evaluate T cell function. An intracellular interferon-gamma assay will be performed by incubating peripheral blood mononuclear cells overnight with an influenza antigen and evaluating the level of an intracellular interferon-y assay will be performed by incubating peripheral blood mononuclear cells overnight with an influenza antigen and evaluating the level of interferon -gamma in activated T cells. Vaccination should increase numbers of T cells producing interferon -gamma. Vaccination should increase numbers of T cells producing interferon -gamma.This evaluation will be done using blood drawn at 5 time points, including pre-vaccination and post vaccination at 2, 4, 12 and 24 weeks.
Measure of antigen specific B cells from pre-vaccination though 24 weeks post-vaccination | 24 weeks
  Measure of antigen specific B cells to determine B cell responsiveness to the pneumococcal vaccine. Polysaccharides from various pathogenic strains will be conjugated to a fluorescent molecule such as fluorescein isothiocyanate (FITC). These constructs will be combined with B cell markers to evaluate pneumococcal specific B cells pre- and post-vaccination. If vaccination is successful, there should be an increase in antigen specific B cells.
Total PnC-IgG, IgG2, PnC-IgG1 and IgG3 levels from pre-vaccination though 24 weeks post-vaccination | 24 weeks
  Total PnC-IgG levels and IgG2 levels will be determined by EIA using commercially available, FDA cleared kits (The Binding Site). PnC-IgG1 and IgG3 levels will be measured by ELISA using commercially available kits that we will modify in-house with optimized reagents for detection of IgG1 and IgG3 isotopes, standardized against a reference serum. This evaluation will be done using blood drawn at 5 time points, including pre-vaccination and post vaccination at 2, 4, 12 and 24 weeks.
Evaluate both FcyRIIa and FcyRIII polymorphisms | up to 24 weeks
  Effectiveness of pneumococcal vaccines has an association with FcyRIIa that is expressed predominantly on phagocytic cells such as neutrophils and macrophages. There are no reports that suggest polymorphisms in FcyRIII are associated with improved efficacy of pneumococcal vaccines. However, therapeutic antibodies for the treatment of cancer such as rituximab have demonstrated that there is a survival advantage of individuals that have the FcyRIIa (H131R) and FcyRIII (V158F) polymorphisms. By evaluating both FcyRIIa and FcyRIII we can position ourselves to evaluate the use of vaccines and therapeutics in cancer.

SECONDARY OUTCOMES:
Assess outcomes of MM patients after vaccination | up to 10 years
  Long term outcomes data will be collected from the medical record of MM patients in order to access the impact of vaccination on health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thompson, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States